CLINICAL TRIAL: NCT04942002
Title: Retrobulbar Methylprednisolone as Adjunctive Treatment in Optic Neuritis. Randomized Controlled Trial.
Brief Title: Retrobulbar Methylprednisolone as Adjunctive Treatment in Optic Neuritis Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neu-21-01
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Optic Neuritis; Treatment; Methylprednisolone
Keywords: Optic Neuritis; Methylprednisolone; Retrobulbar injection
MeSH Terms: conditions — Optic Neuritis | interventions — Methylprednisolone Acetate; Methods

STUDY DESIGN:
Intervention Model Description: Randomized groups (2)
  1. Standard treatment + placebo
  2. Standard treatment + intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants won't be aware to which group they were assigned. Investigator in charge of assessing outcomes and analyzing data won't be aware to which group participants were assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment + placebo (Placebo Comparator): Intravenous Methylprednisolone succinate (1 g daily for 5 days) + paraocular injection of 0.9% saline solution
  Interventions: Drug: Placebo Comparator: Standard treatment + placebo
- Standard treatment + intervention (Experimental): Intravenous Methylprednisolone succinate (1 g daily for 5 days) + retrobulbar injection of 2 cc (40 mg/mL) to methylprednisolone acetate
  Interventions: Drug: Methylprednisolone Acetate 40 MG/ML [Depo-Medrol]

INTERVENTIONS:
Drug: Methylprednisolone Acetate 40 MG/ML [Depo-Medrol] — Retrobulbar injection performed by care provider
  Other Names: Experimental: Standard treatment + intervention
  Arms: Standard treatment + intervention
Drug: Placebo Comparator: Standard treatment + placebo — Intravenous Methylprednisolone succinate (1 g daily for 5 days) + paraocular injection of 0.9% saline solution by care provider
  Other Names: 1. Standard treatment + placebo
  Arms: Standard treatment + placebo

SUMMARY:
A double-blind prospective randomized clinical trial of treatment for optic neuritis comparing visual outcome of patients treated by standard therapy (intravenous methylprednisolone) + placebo injection and standard therapy + retrobulbar methylprednisolone.

DETAILED DESCRIPTION:
A double-blind prospective randomized clinical trial of treatment for optic neuritis comparing visual outcome of patients treated by standard therapy (intravenous methylprednisolone) + placebo injection and standard therapy + retrobulbar methylprednisolone.

Enrollment: 50. Randomized groups (2)

1. Standard treatment + placebo
2. Standard treatment + intervention Masking: Double (participant and outcomes assessor) Participants won't be aware to which group they were assigned. Investigator in charge of assessing outcomes and analyzing data won't be aware to which group participants were assigned

ELIGIBILITY:
Inclusion Criteria:

* Both genres
* Age between 18 and 85 years old.
* Optic neuritis diagnosis ( relative afferent pupillary defect, acquired dyschromatopsia, low vision, prechiasmatic campimetric defect)
* 1 month after symptoms started
* If is a bilateral simultaneous optic neuritis the eye with the worst vision will be included.
* if is a bilateral sequential optic neuritis the eye with lees 1 month evolution will be included.

Exclusion Criteria:

* Visual field better than 20/60 at the beginning of the study.
* History of optic neuritis in the eye under study.
* History of additional ophthalmological or neurological pathology that has caused visual loss in the eye under study.
* History of previous treatment with intravenous methylprednisolone since the onset of symptoms.
* History of high myopia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Visual Capacity | Initial visit, 2-week visit, 1-month visit, 3-month visit
  Best corrected visual acuity

SECONDARY OUTCOMES:
Change from Baseline Color vision | Initial visit, 2-week visit, 1-month visit, 3-month visit
  Color vision as measured by Ishihara plates
Change from Baseline Visual field defect | Initial visit, 2-week visit, 1-month visit, 3-month visit
  Visual fields as measured by Goldmann perimetry
Change from Baseline Oct pRNFL (microns) | 2-week visit, 3-month visit
  Nerve fiber thickness as measured by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cárdenas-Belaunzarán, MD, MSc, Study Director — Asociación Para Evitar la Ceguera en México I.A.P; Karen Flores-Guevara, MD, Principal Investigator — Asociación Para Evitar la Ceguera en México I.A.P
Locations (1):
- Jorge Cárdenas Belaunzarán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
This study is confidential and no information will be shared with the participants.

REFERENCES:
- [Background] Yau GS, Lee JW, Lau PP, Tam VT, Wong WW, Yuen CY. Longitudinal Changes in Retinal Nerve Fibre Layer Thickness after an Isolated Unilateral Retrobulbar Optic Neuritis: 1-Year Results. Neuroophthalmology. 2015 Jan 22;39(1):22-25. doi: 10.3109/01658107.2014.984230. eCollection 2015 Feb. PMID 27928326
- [Background] Prasad S, Volpe NJ, Balcer LJ. Approach to optic neuropathies: clinical update. Neurologist. 2010 Jan;16(1):23-34. doi: 10.1097/NRL.0b013e3181be6fad. PMID 20065793
- [Background] Van Stavern GP. Metabolic, hereditary, traumatic, and neoplastic optic neuropathies. Continuum (Minneap Minn). 2014 Aug;20(4 Neuro-ophthalmology):877-906. doi: 10.1212/01.CON.0000453313.37143.9b. PMID 25099099
- [Background] Costello F. Inflammatory optic neuropathies. Continuum (Minneap Minn). 2014 Aug;20(4 Neuro-ophthalmology):816-37. doi: 10.1212/01.CON.0000453316.60013.52. PMID 25099096
- [Background] Confino E, Mayden KL, Giglia RV, Vermesh M, Gleicher N. Pitfalls in sonographic imaging of the incompetent uterine cervix. Acta Obstet Gynecol Scand. 1986;65(6):593-7. doi: 10.3109/00016348609158394. PMID 3541483
- [Background] Rappoport D, Goldenberg-Cohen N, Luckman J, Leiba H. Parainfectious optic neuritis: manifestations in children vs adults. J Neuroophthalmol. 2014 Jun;34(2):122-9. doi: 10.1097/WNO.0000000000000113. PMID 24667772
- [Background] Boudreault K, Durand ML, Rizzo JF 3rd. Investigation-Directed Approach to Inflammatory Optic Neuropathies. Semin Ophthalmol. 2016;31(1-2):117-30. doi: 10.3109/08820538.2015.1114835. PMID 26959137
- [Background] Bennett JL. Finding NMO: The Evolving Diagnostic Criteria of Neuromyelitis Optica. J Neuroophthalmol. 2016 Sep;36(3):238-45. doi: 10.1097/WNO.0000000000000396. PMID 27529327
- [Background] Abouna GM. Extracorporeal liver perfusion using a new perfusion chamber. Lancet. 1968 Dec 7;2(7580):1216-8. doi: 10.1016/s0140-6736(68)91696-6. No abstract available. PMID 4177207
- [Background] Borvak J, Mayer V. UV-absorbance profile of human leukocytic ultrafiltrate after affinity chromatography on immobilized m-aminophenyl boronic acid: implication for transfer factor purification. Acta Virol. 1985 Mar;29(2):119-28. PMID 2860795
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] Jabs DA, Rosenbaum JT, Foster CS, Holland GN, Jaffe GJ, Louie JS, Nussenblatt RB, Stiehm ER, Tessler H, Van Gelder RN, Whitcup SM, Yocum D. Guidelines for the use of immunosuppressive drugs in patients with ocular inflammatory disorders: recommendations of an expert panel. Am J Ophthalmol. 2000 Oct;130(4):492-513. doi: 10.1016/s0002-9394(00)00659-0. PMID 11024423
- [Background] Jermak CM, Dellacroce JT, Heffez J, Peyman GA. Triamcinolone acetonide in ocular therapeutics. Surv Ophthalmol. 2007 Sep-Oct;52(5):503-22. doi: 10.1016/j.survophthal.2007.06.004. PMID 17719372
- [Background] Arifulin AA, Burenkov MS, Davidenkov AV, Pichugin VIu, Salimov RM. [Mechanism of the effect of nonionizing radiation on animals at the level of sensory systems]. Radiobiologiia. 1986 Mar-Apr;26(2):247-50. Russian. PMID 3704120
- [Background] Rawson MD, Liversedge LA, Goldfarb G. Treatment of acute retrobulbar neuritis with corticotrophin. Lancet. 1966 Nov 12;2(7472):1044-6. doi: 10.1016/s0140-6736(66)92025-3. No abstract available. PMID 4162503
- [Background] Schimek RA, Newsom SR. Restoration of vision in temporal arteritis by retrobulbar injections of steroids. Am J Ophthalmol. 1966 Oct;62(4):693-6. doi: 10.1016/0002-9394(66)92196-9. No abstract available. PMID 5929135
- [Background] Gould ES, Bird AC, Leaver PK, McDonald WI. Treatmenf of optic neuritis by retrobulbar injection of triamcinolone. Br Med J. 1977 Jun 11;1(6075):1495-7. doi: 10.1136/bmj.1.6075.1495. PMID 326332
- [Background] Knudsen LL. Retrobulbar injection of methylprednisolone in diffuse diabetic macular edema. Retina. 2004 Dec;24(6):905-9. doi: 10.1097/00006982-200412000-00010. PMID 15579988
- [Background] Hayashi K, Hayashi H. Intravitreal versus retrobulbar injections of triamcinolone for macular edema associated with branch retinal vein occlusion. Am J Ophthalmol. 2005 Jun;139(6):972-82. doi: 10.1016/j.ajo.2004.12.087. PMID 15953425
- [Background] Bordaberry M, Marques DL, Pereira-Lima JC, Marcon IM, Schmid H. Repeated peribulbar injections of triamcinolone acetonide: a successful and safe treatment for moderate to severe Graves' ophthalmopathy. Acta Ophthalmol. 2009 Feb;87(1):58-64. doi: 10.1111/j.1755-3768.2008.01171.x. Epub 2008 Oct 7. PMID 18937809
- [Background] Boniuk V, Nockowitz R. Perforation of the globe during retrobulbar injection: medicolegal aspects of four cases. Surv Ophthalmol. 1994 Sep-Oct;39(2):141-5. doi: 10.1016/0039-6257(94)90159-7. PMID 7801222
- [Background] Raghava S, Hammond M, Kompella UB. Periocular routes for retinal drug delivery. Expert Opin Drug Deliv. 2004 Nov;1(1):99-114. doi: 10.1517/17425247.1.1.99. PMID 16296723
- [Background] Abel AD, Carlson JA, Bakri S, Meyer DR. Sclerosing lipogranuloma of the orbit after periocular steroid injection. Ophthalmology. 2003 Sep;110(9):1841-5. doi: 10.1016/S0161-6420(03)00560-8. PMID 13129887
- [Background] Parikh S, Shanmugam MP, Biswas J. Bisected macula following retrobulbar steroid injection. Indian J Ophthalmol. 1999 Dec;47(4):247-8. PMID 10892482